CLINICAL TRIAL: NCT03585686
Title: The Prospective Non-randomized Phase II Clinical Trial of Vemurafenib in Combination With Cytarabine and 2-chlorodeoxyadenosine in Children With Langerhans-cell Hisitocytosis With BRAF V600E Mutation
Brief Title: A Combination of Vemurafenib, Cytarabine and 2-chlorodeoxyadenosine in Children With LCH and BRAF V600E Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2017-02
Record Dates: First submitted 2018-07-06; First posted 2018-07-13 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: LCH; Langerhans; histiocytosis; vemurafenib; BRAF
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Histiocytosis | interventions — Vemurafenib; Cytarabine; Cladribine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vemurafenib (Experimental): vemurafenib, Cytarabine, 2-chlorodeoxyadenosine
  Interventions: Drug: Vemurafenib; Drug: Cytarabine; Drug: 2-chlorodeoxyadenosine

INTERVENTIONS:
Drug: Vemurafenib — vemurafenib 20 mg/kg/day
Drug: Cytarabine — 100 mg/m2/12 h, days 1-5
Drug: 2-chlorodeoxyadenosine — 6 mg/m2/d, days 1-5

SUMMARY:
Langerhans cell histiocytosis (LCH) is a disease caused by clonal expansion, proliferation, and dissemination of cells that are phenotypically close to Langerhans cells in different tissues and organs. The clinical presentation of LCH varies greatly from one solid bone tumor to multisystem lesion that involves liver, spleen and bone marrow.

The basis of LCH is the clonal proliferation of the pathological cells. These cells express CD1a and CD207 markers on their surface and originate from myeloid progenitors. The main event in life circle of these cells is the MEK-ERK cascade mutation. The most common mutation is the substitution of valine for glutamic acid in position 600 of BRAF gene. The influence of this mutation was confirmed by G.Badalyan-Very et al. in 2010. About 64% of all LCH are caused by clonal proliferation due to BRAF V600E mutation.

Despite generally good results of therapy of monosystemic LCH, the treatment of LCH with risk organs lesion is still a challenge: 5-years survival is as low as 40-50%.

Combination of cytarabine and 2-chlorodeoxyadenosine was supposed to improve the results, but the cost was a very high toxicity, that limits the application of the regimen in patients with severe infections.

Currently, there is a lot of information on BRAF V600E inhibitors in patients with LCH and other histiocytic disorders. Most of them report the dramatic efficacy of BRAF V600E inhibitors but after quick effect patients usually burden minimal disease activity ("plateau" effect). However, discontinuation of the therapy results in quick disease reactivation.

Considering this a trial that combines targeted therapy (vemurafenib) and low-dose chemotherapy (cytarabine and 2-chlorodeoxyadenosine) in order to achieve complete response with manageable toxicity is proposed.

DETAILED DESCRIPTION:
Langerhans cell histiocytosis (LCH) is a disease caused by clonal expansion, proliferation, and dissemination of cells that are phenotypically close to Langerhans cells to different tissues and organs. The clinical presentation of LCH varies greatly from one solid bone tumor to multisystem lesion that involves liver, spleen and bone marrow.

The basis of LCH is the clonal proliferation of the pathological cells. These cells express CD1a and CD207 markers on their surface and originate from myeloid progenitors. The main event in life circle of these cells is the MEK-ERK cascade mutation. The most common mutation is the substitution of valine for glutamic acid in position 600 of BRAF gene. The influence of this mutation was confirmed by G.Badalyan-Very et al. in 2010. About 64% of all LCH are caused by clonal proliferation due to BRAF V600E mutation.

Despite generally good results of therapy of monosystemic LCH, the treatment of LCH with risk organs lesion is still a challenge: 5-years survival is as low as 40-50%.

Combination of cytarabine and 2-chlorodeoxyadenosine was supposed to improve the results, but the cost was very high toxicity, that limits the application of the regimen in patients with severe infections.

Currently, there is a lot of information on BRAF V600E inhibitors in patients with LCH and other histiocytic disorders. Most of them report the dramatic efficacy of BRAF V600E inhibitors but after quick effect patients usually burden minimal disease activity ("plateau" effect). However, discontinuation of the therapy results in quick disease reactivation.

Considering this a trial that combines targeted therapy (vemurafenib) and low-dose chemotherapy (cytarabine and 2-chlorodeoxyadenosine) in order to achieve complete response with manageable toxicity is proposed.

Patients who met the eligibility criteria evaluate their condition using DAS score on Day 0 and start the therapy with oral intake of vemurafenib 20 mg/kg/d rounded off to a whole capsule from day 1 to day 28. NB! In life-threatening cases, the treatment can be started empirically, without BRAF V600E detection in any affected tissue.

During that period their condition will be strictly monitored in order to control BRAF V600E inhibitor side effects. Moreover, serum levels of vemurafenib should be evaluated on any two points after day 3 and before day 28. Serum concentration should be measured with the mass-spectrometry method in the positive ionization regimen.

On day 28 condition must be evaluated with DAS again and vemurafenib intake should be stopped. On day 29, Ara-C + 2-CdA course №1 should be started. It takes 5 days, on day 34 vemurafenib intake should be continued.

Each patient should undergo 3 courses of Ara-C + 2-CdA with 28 days between each course. After each course, G-CSF stimulation and proper antibacterial/antifungal therapy are to be applied.

Before each course, patients condition should be evaluated with DAS scale. After Ara-C + 2-CdA, №3 patient should undergo a more thorough evaluation that includes bone marrow aspiration. After that vemurafenib intake should be stopped and mono 2-CdA course starts. After 5 days of the course, vemurafenib intake shouldn't be restarted.

After 3 courses of mono 2-CdA, all specific therapy stops. On each DAS evaluation point, serum for digital droplet polymerase chain reaction (ddPCR) should also be collected. With the help of ddPCR, it could be possible to analyze cell-free DNA (cfDNA) harboring BRAF V600E mutation and thus to create a method of disease activity control.

Taking into account the small potential number of the included patients the analysis of data will be based on Simon two-step design.

All reactivation-free survival and overall survival rates will be evaluated with standard Kaplan-Mayer method.

All severe side effects will be evaluated with standard CTCAE scale.

All operations with patients' data, informed consents will be performed according to the internal SOPs.

ELIGIBILITY:
Inclusion Criteria:

* 0-18 years old
* histologically verified diagnosis of LCH (CD1a+/CD207+)
* verified BRAF V600E mutation in the biopsy specimen AND/OR CD34+ isolate (NB! In life-threatening cases, vemurafenib can be administered BEFORE BRAF V600E mutation confirmation. It's recommended to stop vemurafenib therapy if no clinically significant positive dynamic was achieved after 7 days of intake)
* QTc < 0.5 s
* no previously documented cardiac diseases
* signed informed consent

Exclusion Criteria:

* withdrawal of informed consent
* QTc > 0.5 s or long QT syndrome
* use of antiarrhythmic medication
* persistent electrolytic disorders

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-06-26 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The overall response rate (ORR) proportion | 16 weeks
  ORR is the sum of complete response rate (CRR) and partial response rate (PRR) which define as DAS score 0-1 and 2-3 respectfully.

SECONDARY OUTCOMES:
The reactivation/progression free survival | 1 year
  RFS is a time from the therapy start to reactivation, progression or death due to any cause or to last evaluation up to the time of analysis. Analysis will be made with Kaplan-Mayer method with 95% confidence interval.
The proportion of of patients with severe adverse effects | 30 days
  The proportion of of patients with severe adverse effects of therapy according to CTCAE (ver 4.0)
Overall survival | 2 years
  OS is a time from the therapy start to death due to any cause or to the last evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Evseev D, Osipova D, Kalinina I, Raykina E, Ignatova A, Lyudovskikh E, Baidildina D, Popov A, Zhogov V, Semchenkova A, Litvin E, Kotskaya N, Cherniak E, Voronin K, Burtsev E, Bronin G, Vlasova I, Purbueva B, Fink O, Pristanskova E, Dzhukaeva I, Erega E, Novichkova G, Maschan A, Maschan M. Vemurafenib combined with cladribine and cytarabine results in durable remission of pediatric BRAF V600E-positive LCH. Blood Adv. 2023 Sep 26;7(18):5246-5257. doi: 10.1182/bloodadvances.2022009067. PMID 37216396